CLINICAL TRIAL: NCT00747708
Title: Randomised Control Trial to Compare the Effects of G-CSF and Autologous Bone Marrow Progenitor Cells Infusion on the Quality of Life and Left Ventricular Function in Patients With Heart Failure Secondary to Ischaemic Heart Disease
Brief Title: Bone Marrow Derived Adult Stem Cells for Chronic Heart Failure
Acronym: REGEN-IHD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Anthony Mathur, Lead Cardiologist, Barts & The London NHS Trust
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 04/Q0603/13; 2005-002706-27 (EudraCT)
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Ischaemic Heart Failure
Keywords: heart failure; coronary heart disease; adult stem cells; bone marrow progenitor cells; bone marrow stem cells; autologous; granulocyte-colony stimulating factor; left ventricular function; intracoronary injection; intramyocardial injection
MeSH Terms: conditions — Heart Failure; Coronary Disease | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peripheral (Experimental): Patients are randomised in a 1:1 ratio to receive granulocyte-colony stimulating factor (G-CSF) or placebo injection
  Interventions: Drug: Granulocyte-colony stimulating factor
- Percutaneous intracoronary injection (Experimental): All patients will receive granulocyte-colony stimulating factor injections followed by a bone marrow aspiration. Patients will be randomised in a 1:1 ratio to receive intracoronary injections of bone marrow derived stem/progenitor cells or placebo infusion through a percutaneous route
  Interventions: Drug: Granulocyte-colony stimulating factor; Procedure: Percutaneous intracoronary injection
- Percutaneous intramyocardial injection (Experimental): All patients will receive granulocyte-colony stimulating factor injections followed by a bone marrow aspiration. Patients will be randomised in a 1:1 ratio to receive intramyocardial injections of bone marrow derived stem/progenitor cells or placebo infusion through a percutaneous route
  Interventions: Drug: Granulocyte-colony stimulating factor; Procedure: Percutaneous intramyocardial injection

INTERVENTIONS:
Drug: Granulocyte-colony stimulating factor — 5 days subcutaneous injection
  Other Names: G-CSF
Procedure: Percutaneous intracoronary injection — Bone marrow derived stem/progenitor cells or placebo infusion is delivered through an over-the-wire balloon catheter into the target coronary vessels using a stop-flow technique.
  Arms: Percutaneous intracoronary injection
Procedure: Percutaneous intramyocardial injection — Direct intramyocardial injections of bone marrow derived stem/progenitor cells or placebo will be delivered using the electromechanical NOGA mapping and injection system
  Arms: Percutaneous intramyocardial injection

SUMMARY:
The purpose of this study is to determine whether adult bone marrow derived stem/progenitor cells improve cardiac function and symptoms in patients with heart failure and to establish the optimal method of delivery of these cells.

Study hypotheses:

* Administration of G-CSF to patients with heart failure secondary to ischaemic heart disease will lead to an increase in circulating progenitor cells as measured by peripheral CD34+ positive cell counts
* Cardiac function and symptoms will improve in patients in whom the peripheral CD34+ counts increase in response to G-CSF administration
* Direct coronary injection of autologous bone marrow derived stem cells will confer an additional improvement in cardiac function and symptoms above that derived from G-CSF infusion alone
* Direct intramyocardial injection of autologous bone marrow derived stem cells will lead to an improvement in cardiac function and symptoms above that derived from G-CSF infusion alone

DETAILED DESCRIPTION:
The study involves three arms that compare the method of autologous bone marrow cel administration in patients with chronic heart failure. Each arm has a comparative group that contains either saline injection (peripheral arm that injects GCSF alone) or serum (the two interventional arms-intracoronary and intramyocardial injection).

The protocol (on the advice of the ethics committee) is divided into a 58 patients pilot study followed by recruitment into the intramyocardial arm (30 patients randomised 1:1 cells in serum vs serum alone) and then recruitment into the intracoronary and peripheral arms (30 patients randomised 1:1 cells in serum vs serum alone in each arm).

The study has been powered around the use of advanced imaging to measure within group changes in ejection fraction at 12 months as the primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with a diagnosis of heart failure secondary to ischaemic heart disease who are on optimal heart failure treatment and no further treatment options available
* Patient has been considered for an implantable defibrillator in keeping with NICE guidelines

Exclusion Criteria:

* Recent acute coronary syndrome as judged by a rise of Troponin above normal values in the last 6 months
* The presence of cardiogenic shock
* The presence of acute left and/or right-sided pump failure as judged by the presence of pulmonary oedema and/or new peripheral oedema
* Known severe pre-existent left ventricular dysfunction (ejection fraction < 10% prior to randomisation)
* Congenital cardiac disease
* Cardiomyopathy secondary to a reversible cause e.g. thyroid disease, alcohol abuse, hypophosphataemia, hypocalcaemia, cocaine abuse, selenium toxicity & chronic uncontrolled tachycardia
* Cardiomyopathy in association with a neuromuscular disorder e.g. Duchenne's progressive muscular dystrophy
* Contra-indication for bone marrow aspiration
* Known active infection
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) syphilis or HTLV
* Lifestyle with high risk for infection with HIV, HBV or HCV syphilis or HTLV
* Serum creatinine >200 umol/L
* Chronic inflammatory disease
* Serious known concomitant disease with a life expectancy of less than one year
* Follow-up impossible (no fixed abode, etc)
* Previous participation in this study
* Female subjects of childbearing potential
* Atrial fibrillation
* Patients who have responded to the implantation of a biventricular pacemaker
* Weight >140kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-08; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in global left ventricular ejection fraction | 12 months

SECONDARY OUTCOMES:
Change in quality of life | 6 months
Occurence of major adverse cardiac event | 12 months
Change in quality of life | 12 months
Change in NT-proBNP | 6 months
change in NYHA class | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, FRCP FESC Ph, Principal Investigator — Barts and the London NHS Trust
Locations (1):
- London Chest Hospital, Barts and the London NHS Trust, London, London, United Kingdom